CLINICAL TRIAL: NCT02782325
Title: Safety and Efficacy of Fecal Microbiome Transplantation (FMT) in the Treatment of Antibiotic Dependent Pouchitis (ADP)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due low efficacy of FMT in interim analysis.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: OpenBiome (Industry); Crohn's and Colitis Foundation (Other); The Broad Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-1310; FMTADP (Other: UNC-CH)
Record Dates: First submitted 2016-05-12; First posted 2016-05-25 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2018-12

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active FMT, then open label FMT (Active Comparator): Endoscopic application of OpenBiome FMT Lower Delivery followed by 2 weeks of treatment with OpenBiome FMT Capsules G3 with follow-up at week 4, 8, 16 and 24 after inclusion. In case the study patient does not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study he/she will be offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an additional endoscopic FMT followed by 2 weeks of oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
  Interventions: Biological: Active FMT, then open label FMT
- Placebo FMT, then open label FMT (Placebo Comparator): Endoscopic application of Placebo FMT Lower Delivery followed by 2 weeks of treatment with Placebo FMT Capsules G3 with follow-up at week 4, 8, 16 and 24 after inclusion. In case the study patient does not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study he/she will be offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an additional endoscopic FMT followed by 2 weeks of oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
  Interventions: Biological: Placebo FMT, then open label FMT

INTERVENTIONS:
Biological: Active FMT, then open label FMT — Endoscopic application of OpenBiome FMT Lower Delivery followed by 2 weeks of treatment with OpenBiome FMT Capsules G3 with follow-up at week 4, 8, 16 and 24 after inclusion. In case the study patient does not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study he/she will be offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an additional endoscopic FMT followed by 2 weeks of oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
  Other Names: Active FMT
  Arms: Active FMT, then open label FMT
Biological: Placebo FMT, then open label FMT — Endoscopic application of Placebo FMT Lower Delivery followed by 2 weeks of treatment with Placebo FMT Capsules G3 with follow-up at week 4, 8, 16 and 24 after inclusion. In case the study patient does not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study he/she will be offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an additional endoscopic FMT followed by 2 weeks of oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
  Other Names: Placebo FMT
  Arms: Placebo FMT, then open label FMT

SUMMARY:
Antibiotic dependent pouchitis (ADP) is predestined to benefit from FMT, since bacterial dysbiosis, which can only be controlled with antibiotics, appears to be the major driver of the clinical symptoms. This is a proof of concept randomized placebo controlled trial, in which 50% of the patients will receive FMT and 50% will receive a placebo FMT. Additionally the trial offers an open label extension period.

DETAILED DESCRIPTION:
FMT for ADP is a promising approach, given the documented role of bacteria in the pathogenesis. In contrast to patients with C. difficile colitis, in whom a single FMT is highly effective, in patients with Inflammatory Bowel Disease (IBD) an intensified therapy with daily or repeated FMT may be more beneficial. Whereas repeated endoscopic application are not feasible and repeated enema applications are not favored by patients a combination of endoscopic FMT and consecutive maintenance therapy with oral FMT using the FMT capsule G3 produced by OpenBiome to help establish the donor microbiome in the host seems to be the most promising approach. The objective of this trial is to evaluate the safety of FMT in patients with ADP and to estimate the effect size to be achieved from FMT therapy in patients with ADP for subsequent evaluation in a large definitive trial. A secondary objective is to study the microbial engraftment of donor FMT in the recipients.

This proof of concept randomized placebo controlled trial with an open label extension period will evaluate the safety and efficacy of an initial endoscopic FMT followed by 14 days of oral FMT. The study has two distinct outcomes, a clinical and translational aim, to investigate the effect of FMT in patients with ADP.

Aim1: Evaluation of safety, tolerability and clinical effectiveness (measured as clinical response or remission and discontinuation of antibiotic therapy) of FMT in patients with ADP.

Aim 2: Evaluation of the impact of FMT on the fecal bacterial microbiome in patients with ADP, which will provide functional data about possible mechanisms of this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Man or woman between 18 and 70 years of age.
* Ileal Pouch-Anal Anastomosis (IPAA) after colectomy for ulcerative colitis
* Active pouchitis, defined as a modified pouch disease activity index (mPDAI) ≥ 5 and a history of ≥ 4 antibiotic therapies for pouchitis in the last 12 months

or

- Need for ongoing antibiotic therapy (> 4 weeks) to maintain clinical remission and a history of at least 2 attempts in the last 24 months to stop antibiotic therapy resulting in pouchitis episodes.

Exclusion Criteria:

* Treatment with biologics (e.g. infliximab, adalimumab, golimumab, vedolizumab)
* Treatment with immunomodulators (azathioprine, 6-mercaptopurine (6-MP), methotrexate), steroids or any investigational drugs
* Use of cholestyramine
* Crohn's disease of the pouch
* Known cytomegalovirus infection of the pouch
* Clostridium difficile infection
* Isolated cuffitis
* Clinical significant strictures of the pouch inlet or outlet
* Concurrent intestinal obstruction
* History of familial adenomatous polyposis
* History of uncontrolled lactose intolerance
* History of confirmed (serological test and/or histology) celiac disease
* Pregnancy, breast feeding, or planning to become pregnant during the trial
* Non - steroidal inflammatory medications (NSAIDs) as long-term treatment, defined as use for at least 4 days a week each month
* Dysphagia (oropharyngeal, esophageal, functional, neuromuscular)
* History of recurrent aspiration episodes
* Proven Gastroparesis
* Allergy to the following generally regarded as safe ingredients (GRAS): glycerol, acid resistant hypromellose (HPMC), gellan gum, cocoa butter, titanium dioxide
* Adverse event attributable to previous FMT
* Allergy/intolerance to pump inhibitor therapy
* Any condition for which the investigator thinks the FMT treatment may pose a health risk (e.g. severely immunocompromised)
* Participation in another clinical trial within the last 30 days, simultaneous participation in another clinical trial, or previous participation in this trial
* During the trial period until one week after the trial end: Non-use of appropriate contraceptives in females of childbearing potential (e.g. condoms, intrauterine device (IUD), hormonal contraception, or other means considered adequate by the responsible investigator) or in males with a child-fathering potential (condoms, or other means considered adequate by the responsible investigator during treatment - Well-founded doubt about the patient's cooperation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Herfarth, MD, PhD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The final results of the trial will be posted on clinical trials.gov. No individual patient data will be posted.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient after screening since he met an exclusion criterion. 6 patients went on to randomization
Groups:
- Open Label FMT Period: Participants who do not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study were offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an open label endoscopic FMT followed by 2 weeks of open label oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
Period: Blinded FMT Treatment (up to 24 Weeks)
Arm/Group | Active FMT, Then Open Label FMT | Placebo FMT, Then Open Label FMT | Open Label FMT Period
Started | 4 | 2 | 0
Completed | 0 | 0 | 0
Not Completed | 4 | 2 | 0
Not completed — Lack of Efficacy | 4 | 2 | 0
Period: Open Label FMT Period (up to 24 Weeks)
Arm/Group | Active FMT, Then Open Label FMT | Placebo FMT, Then Open Label FMT | Open Label FMT Period
Started (One patient declined participation in the open label extension arm) | 0 | 0 | 5 (1 participant decided to not participate in the open label period)
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active FMT, Then Open Label FMT | Placebo FMT, Then Open Label FMT | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With FMT Related Adverse Event
Description: Number of patients with FMT related adverse event (classified according to MedDRA; lowest level term) and categorized according to CTCAE Version 4.0. The safety was assessed in the randomized placebo controlled segment of the study over 24 weeks after initial endoscopic FMT weeks and if the patient should enter the open label extension part of the study also for 24 weeks after initial open label FMT. 6 patients participated in the randomized arm and 5 patients in the open label extension arm.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Phase: Active FMT: Endoscopic application of OpenBiome FMT Lower Delivery followed by 2 weeks of treatment with OpenBiome FMT Capsules G3 with follow-up at week 4, 8, 16 and 24 after inclusion. In case the study patient does not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study he/she will be offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an additional endoscopic FMT followed by 2 weeks of oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
- Randomized Phase: Placebo: Endoscopic application of Placebo FMT Lower Delivery followed by 2 weeks of treatment with Placebo FMT Capsules G3 with follow-up at week 4, 8, 16 and 24 after inclusion. In case the study patient does not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study he/she will be offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an additional endoscopic FMT followed by 2 weeks of oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
- Open Label FMT: Participants who do not achieve clinical remission at week 4 or experiences a flare of disease on day 15-28 after start of the study were offered the possibility to participate in open label extension after at least 10 day of antibiotic therapy with an open label endoscopic FMT followed by 2 weeks of open label oral FMT. Follow-up will occur in open label at week 4, 8, 16 and 24 after open label FMT.
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
Number analyzed (Participants) | 4 | 2 | 5
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Patients in Clinical Remission Week 4 After Endoscopic and Oral FMT
Description: Clinical remission as defined by a composite assessment, of which all criteria need to be met: Clinical modified pouch diseases activity index (mPDAI) score ≤4 points and no need for antibiotic therapy at week 4.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
Number analyzed (Participants) | 4 | 2 | 5
Participants | 0 | 0 | 1

3. Secondary Outcome: Number of Patients in Clinical Remission Week 16
Description: Clinical remission as defined by a composite assessment, of which all criteria need to be met: Clinical mPDAI score ≤4 points and no need for antibiotic therapy at week 16.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
Number analyzed (Participants) | 4 | 2 | 5
Participants | 0 | 0 | 1

4. Secondary Outcome: Number of Patients With Endoscopic Improvement Week 4 After Endoscopic and Oral FMT
Description: Endoscopic improvement of active pouchitis (decrease from baseline in modified pouch disease activity index endoscopic subscore > 2 points) at week 4.
Time Frame: 4 weeks
Population: None of the patients in the randomized phase underwent an endoscopy at week 4 since they all relapsed before week 4. In the open label extension only 1 patient underwent endoscopy at week 4 and the pouch was endoscopically unchanged.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
Number analyzed (Participants) | 0 | 0 | 1
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Clinical Response at Week 4 in Patients Entering the Trial With Active Pouchitis Symptoms
Description: This outcome measure is for patients with active pouchitis symptoms entering the trial. Since all patients entered with inactive pouchitis no patient could be evaluated for this outcome.
  Response as defined by a composite assessment of which both criteria has to be met: Decrease from baseline mPDAI clinical subscore > 2 points and no need for antibiotic therapy at week 4.
Time Frame: 4 weeks
Population: Since all patients entered with inactive pouchitis no patient could be evaluated for this outcome.
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Clinical Response Week 8 and Active Pouchitis at Baseline
Description: Response as defined by a composite assessment of which both criteria has to be met: Decrease from baseline mPDAI clinical subscore > 2 points and no need for antibiotic therapy at week 8 of the randomized phase.
Time Frame: 8 weeks
Population: Only 1 patient in the open label FMT completed the week 8 visit, but entered the trial in remission and thus did n to meet the criterion of a decrease of the clinical PDA sub core decrease
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
Number analyzed (Participants) | 0 | 0 | 1
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Patients With Clinical Response i at Week 16 and Active Pouchitis at Baseline
Description: This outcome measure is for patients with active pouchitis symptoms entering the trial. Response as defined by a composite assessment of which both criteria has to be met: Decrease from baseline mPDAI clinical subscore > 2 points and no need for antibiotic therapy at week 16.
Time Frame: 16 weeks
Population: None of the patients in the trial entered the study with symptoms of active pouchitis
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event were collected for 24 weeks after endoscopic FMT in the randomized phase. If patient the patient participated in the open label extension study period adverse events were collected for 24 weeks after endoscopic FMT in the open label extension phase.
Arm/Group | Randomized Phase: Active FMT | Randomized Phase: Placebo | Open Label FMT
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Phase: Active FMT (N=4) | Randomized Phase: Placebo (N=2) | Open Label FMT (N=5)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Urgency (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to the small sample size only exploratory analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT02782325/Prot_SAP_000.pdf